CLINICAL TRIAL: NCT01638715
Title: A Randomized, Multi-Center Biomarker Trial to Predict Therapeutic Responses of Patients With Rheumatoid Arthritis to a Specific Biologic Mode of Action
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Daniel Aletaha, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIOBIO Study; 2012-000139-21 (EudraCT Number)
Record Dates: First submitted 2012-07-03; First posted 2012-07-12 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Biologic therapies; Biomarker; Mode of Action
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Abatacept; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Infliximab (Experimental): Infliximab (Remicade®) will be administered i.v.at a dose of 3 mg/kg at 0 and 2 weeks, and 5 mg/kg at weeks 6, 14, and 22, 30, 38, and 46.
  Interventions: Drug: Remicade
- Abatacept (Experimental): Abatacept (Orencia®) will be given i.v. at weeks 0, 2, 4, and then every 4 weeks until week 48 at a weight adjusted dose: <60 kg Body weight (BW): 500 mg; >60-100 kg BW: 750 mg; alternatively, based on preference and shared decision between patient and physician, patients randomized to the abatacept arm may receive s.c.application at a dose of 125mg weekly.
  Interventions: Drug: Orencia
- Tocilizumab (Experimental): Tocilizumab (Ro-Actemra®) will be administered every 4 weeks at a dose of 8 mg/kg BW (maximum dose of 800 mg); The employed dosage will be calculated using manufacturer guidelines; alternatively, based on preference and shared decision between patient and physician, patients randomized to the tocilizumab arm may receive s.c. application at a dose of 162mg every week.
  Interventions: Drug: Ro-Actemra
- Rituximab (Experimental): Rituximab (Mabthera®) will be given as 1000mg at weeks 0 and 2, and then repeated at weeks 24 and 26. Patients will receive 100 mg methylprednisolon i.v. before each infusion, as well as 1000mg paracetamol, as well as 50mg diphenhydramine hydrochloride (Dibondrin©).
  Interventions: Drug: Mabthera

INTERVENTIONS:
Drug: Remicade — - Infliximab (Remicade®) will be administered i.v. at a dose of 3 mg/kg at 0 and 2 weeks, and 5 mg/kg at weeks 6, 14, and 22, 30, 38, and 46.
  Arms: Infliximab
Drug: Orencia — - Abatacept (Orencia®) will be given i.v. at weeks 0, 2, 4, and then every 4 weeks until week 48 at a weight adjusted dose: <60 kg Body weight (BW): 500 mg; >60-100 kg BW: 750 mg; alternatively, based on preference and shared decision between patient and physician, patients randomized to the abatacept arm may receive s.c. application at a dose of 125mg weekly.
  Arms: Abatacept
Drug: Ro-Actemra — - Tocilizumab (Ro-Actemra®) will be administered every 4 weeks at a dose of 8 mg/kg BW (maximum dose of 800 mg); The employed dosage will be calculated using manufacturer guidelines; alternatively, based on preference and shared decision between patient and physician, patients randomized to the tocilizumab arm may receive s.c. application at a dose of 162mg every week.
  Arms: Tocilizumab
Drug: Mabthera — - Rituximab (Mabthera®) will be given as 1000mg at weeks 0 and 2, and then repeated at weeks 24 and 26.
  Patients will receive 100 mg methylprednisolon i.v. before each infusion, as well as 1000mg paracetamol, as well as 50mg diphenhydramine hydrochloride (Dibondrin©).
  Arms: Rituximab

SUMMARY:
The purpose of this study is to find biological response patterns of patients with rheumatoid arthritis to drugs with different biologic modes of action. This study should help to predict therapeutic responses and to find the right therapy for the right patient.

DETAILED DESCRIPTION:
The investigators propose a randomised, multi-centre strategic biomarker trial of rheumatoid arthritis (RA) patients with failure to methotrexate or leflunomide to one of the four current biological modes of action: targeting TNF (infliximab); co-stimulation (abatacept); IL-6R (tocilizumab); and B cells (rituximab); all agents are licensed for RA and have evidence for efficacy in this indication. Predictors of response to therapy after 24 weeks will be analysed, and include baseline and follow up assessments of clinical, functional, structural, laboratory tests (routine, autoantibodies, cytokines, gene expression, and susceptibility genes). In a second phase, patients not achieving LDA/REM will be randomised to one of the remaining MoA. Two hundred patients, who are started on a new biological therapy will be enrolled over an estimated period of 5 years; 50 patients per group will be included, and studied for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ≥18 and ≤75 years of age, capable of understanding and signing an informed consent.
2. Classifiable RA according to the 2010 ACR/EULAR criteria (American College of Rheumatology/European League Against Rheumatism classification criteria) or 1987 ARA criteria (Criteria of American Rheumatology Association) (present or past) (2;3)
3. Duration of RA ≤3 years
4. Ongoing conventional DMARD therapy (Disease Modifying Antirheumatic Drugs) with methotrexate (at least 20mg/week, or lower if not tolerated in higher doses) or leflunomide (≥100mg/week), for ≥6 months or ≥3 months with documented worsening of disease activity.
5. Clinical Disease Activity Index (CDAI)≥15 corresponding to moderate to severe disease activity.

Exclusion Criteria:

1. Be incapacitated, largely or wholly bedridden, or confined to a wheelchair, or have little or no ability for self care.
2. Weigh more than 100 kg
3. Use glucocorticoids >10 mg/day prednisone or equivalent
4. Have previously received other treatments for their rheumatic disease:

   1. intra-muscular or intra-articular injection of steroids in the previous month.
   2. monoclonal antibodies or antibody fragments, licenced or investigational
   3. any investigational drug within 3 months prior to screening or within 5 half-lives of the investigational agent, whichever is longer.
   4. Azathioprine or other cytostatic drugs.
5. Have a history of receiving human/murine recombinant products or a known allergy to murine products.
6. Have documentation of seropositivity for human immunodeficiency virus (HIV), or a positive test for hepatitis B surface antigen or hepatitis C ¬antibodies.
7. Have hypergammaglobulinemia
8. Have a history of alcohol or substance abuse within the preceding 6 months.
9. Have or have had a known history of

   1. serious infections (such as, but not limited to hepatitis, pneumonia, or pyelonephritis) in the previous 3 months.
   2. opportunistic infections (eg, herpes zoster, cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 12 months prior to screening.
   3. a chronic or recurrent infectious disease (eg, chronic renal infection, chronic chest infection, COPD, sinusitis, recurrent urinary tract infection, open, draining or infected skin wound or ulcer etc.).
10. Have undergone any joint replacement surgery.
11. Be men and women of childbearing potential without use of adequate birth control measures (e.g., abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, implantable or injectable contraceptives or surgical sterilization), and willingness to continue this precaution for the duration of the study until 6 months after receiving the last medication.
12. Be considered ineligible according to the tuberculosis (TB) eligibility assessment and screening, or show a positive test for latent Tbc using Quantiferon assay, unless treatment with INH has been installed for at least 2 weeks prior to starting trial drug.
13. Show evidence of malignancy, or lymphoproliferative disease, or any history of malignancy within the previous 5 years, with the exception of basal cell or squamous cell carcinoma of the skin that has been fully excised with no evidence of recurrence.
14. Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
15. Be unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access.
16. Have presence of a transplanted solid organ (with the exception of a corneal transplant > 3 months prior to screening).
17. Have a concomitant diagnosis or history of congestive heart failure (New York Heart Association - NYHA - class III or IV) or diverticulitis.
18. Have a known history of a demyelinating disease, such as multiple sclerosis.
19. Be women who are pregnant, nursing, or planning pregnancy within 6 months after the last infusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2012-05; Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Absolute Change in the Simplified Disease Activity Index (SDAI) | 24 Weeks

SECONDARY OUTCOMES:
Relative Change in the SDAI in percent | 24 Weeks
Absolute and relative change in the Clinical Disease Activity Index (CDAI) in percent | 24 Weeks
Absolute and relative change in the Disease Activity Score 28 (DAS28) in percent | 24 weeks
Achieving an SDAI or CDAI response (50%, 70%, 85%) | 24 Weeks
Achieving a EULAR response (European League Against Rheumatism) | 24 Weeks
Achieving an ACR response (20%, 50%, 70%) (American College of Rheumatology) | 24 Weeks
Change in quality of life (EuroQoL-5D, SF-36) | 24 weeks
Change in fatigue (Fatigue Score on the Visual Analog Scale) | 24 Weeks
Proportion achieving a low disease activity state (SDAI ≤11) | 24 Weeks
Proportion achieving a remission state (SDAI ≤3.3) | 24 Weeks
Radiographic progression - (Van der Heijde/Sharp Score) | 6 months and 12 months
Change in physical function (HAQ) | 24 Weeks
Change in sleep (Sleep Score on the Visual Analog Scale) | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Aletaha, MD, Study Director — Medical University of Vienna
Locations (9):
- Austria (6):
  - Gesundheitszentrum Mariahilf, Vienna
  - AKH Wien, Vienna
  - Krankenhaus Hietzing, Vienna
  - Hanusch Krankenhaus, Vienna
  - Wilhelminenspital, Vienna
  - Ordination Wels (Private Medical Office), Wels
- Institute of Rheumatology, Prague, Czechia
- V. A. Nasonova Research Institute of Rheumatology, Moscow, Russia
- Kantonsspital St.Gallen, Klinik für Rheumatologie, Sankt Gallen, Switzerland

REFERENCES:
- [Derived] Studenic P, Bond G, Kerschbaumer A, Becede M, Pavelka K, Karateev D, Stieger J, Puchner R, Mueller RB, Puchhammer-Stockl E, Durechova M, Loiskandl M, Perkmann T, Olejarova M, Luchikhina E, Steiner CW, Bonelli M, Smolen JS, Aletaha D. Torque Teno Virus quantification for monitoring of immunomodulation with biologic compounds in the treatment of rheumatoid arthritis. Rheumatology (Oxford). 2022 Jul 6;61(7):2815-2825. doi: 10.1093/rheumatology/keab839. PMID 34792562